CLINICAL TRIAL: NCT04030689
Title: "Au Labo Sans Ordo ": A 12 Month Local Experimentation of Free HIV Testing Without Prescription in Private Medical and Biological Laboratories in Paris and in the Alpes-Maritimes
Brief Title: Free HIV Testing in Private Biological Laboratories: A New Offer to Encourage HIV Testing
Acronym: ALSO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 19-PP-11
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2019-07

CONDITIONS: HIV Seropositivity; HIV Testing
Keywords: HIV Testing; Combined HIV prevention; Linkage to care; Implementation plan; Cost-effectiveness
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Axis 2: Each patient diagnosed HIV positive following VihTest test will be invited to participate to ALSO-Parcours; This program aimed to decribe the link to care for this population and to make a descriptive analysis of this HIV+ patients.
  Interventions: Other: data collected from patient file

INTERVENTIONS:
Other: data collected from patient file — socio-demographics, previous HIV testing history, history of HIV contamination, clinics HIV related data will be collected for each patient who notified his non-objection to participate to this non interventional study.

SUMMARY:
The program " Au labo sans ordo " aims to increase HIV testing coverage, in order to improve the first stage of the HIV care cascade in Paris and the Alpes-Maritimes, areas facing a much higher HIV epidemic than the other regions in metropolitan France. Both departments are engaged in the Fast Track Cities Initiative.

DETAILED DESCRIPTION:
The program relies on the hypothesis that the opportunity to get tested for HIV for free (called VihTest) in any Private Laboratory (PL), without prior appointment nor prescription, combined with an intense targeted promotion and communication strategy, will significantly increase the testing coverage. This offer might remove some of the multiple barriers to HIV testing and ease the move to action, in particular within key affected populations which contribute to the largest part of the epidemic dynamic.

This program offers a new access to HIV testing. It is developed jointly by local authorities, the health insurance and state regional health agencies, in response to the very low increase of HIV testing coverage despite a diversification of the testing supply and national recommendations for generalized and repeated HIV testing within key populations.

The experimentation will be implemented for 12 months in all Private Laboratories in Paris (164) and the Alpes-Maritimes (107), targeting a 15% increase in the total volume of tests performed outside of hospital settings.

The evaluation process will focus on:

Axis 1 : The number of tests performed and the number of new HIV diagnosis considering the potential substitution effect towards the current testing provision through CeGIDD (free Centers for Information, Diagnosis and Testing) and community-based outreach testing programs.

Axis 2 : The linkage to care following an HIV positive test will be organized and documented and the characteristic of HIV+ population diagnosed after VihTest will be describe (ALSO_PARCOURS) Axis 3: The characteristics of the program's users will be collected and compared 1) to those of PL attendants with a medical prescription for an HIV test and 2) to CeGIDD clients.

Axis 4: The feasibility and acceptability of the program by the PL's staff will be documented using detailed qualitative questionnaire; Axis 5: The cost-effectiveness of scaling-up such a testing strategy and its budgetary impact will be assessed through a microcoasting evalutation.

ELIGIBILITY:
Axis 2

Inclusion Criteria:

* Major
* being diagnosed HIV positive after a VihTest

Exclusion Criteria:

* Minor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Axis 2 Major patient diagnosed HIV positive after a VihTest in a Private Laboratory in Paris or in the Alpes Maritimes.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Positive VihTest | 548 days
  Number of patients enrolled in the study with demographics, risk factors, clinical therapeutic and biological characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Pascal PUGLIESE, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- Hopital l'Archet Service Infectiologie, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided